CLINICAL TRIAL: NCT06401057
Title: Register for Longitudinal Recording of Brain Function in Patients With Brain Diseases
Brief Title: Register for Longitudinal Recording of Brain Function
Status: Recruiting | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Schwendner Maximilian, Principal Investigator, University Hospital Heidelberg
Other Study IDs: Fun-Reg
Record Dates: First submitted 2024-01-07; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Patients With Brain Masses/Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational register study is to establish a registry that completely records and compiles the data from routinely performed technical examinations (navigated transcranial magnetic stimulation, intraoperative neuromonitoring and stimulation, MRI imaging including tractography and connectome) and clinical tests over time (pre-, intra- and postoperative, under adjuvant therapy, as part of follow-up care) of patients with intracranial masses and lesions.

ELIGIBILITY:
Inclusion Criteria:

* Intracranial lesion
* Age ≥ 18 years
* Written consent to participate in the study

Exclusion Criteria:

* Age < 18 years
* Patients not able to give consent
* Patients with intracranial ferromagnetic metal implants
* Patients with implanted electronic devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with brain masses/lesions (especially tumors (cerebral and non-cerebral, inflammation (infectious and non-infectious), vascular pathologies)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive status | until last patient FU up to 48 months
  Higher cognitive functions - determined by the Montreal Cognitive Assessment (MocA)
Language status | until last patient FU up to 48 months
  Language function tested by the Aphasia Check List
Motor status | until last patient FU up to 48 months
  Motor function according to the BMRC scale
cortical data | until last patient FU up to 48 months
  cortical nTMS-Data - distribution according the cortical parellation system
Fiber tracts | until last patient FU up to 48 months
  Volume of fiber tracts
Fiber tracts | until last patient FU up to 48 months
  fractional anisotropy of fiber tracts
structural imaging (Connectome) | until last patient FU up to 48 months
  characteristics of Connectome and Disconnectome analysis (Global Efficiency value)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery Heidelberg University Hospital, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
For selected subgroups, data sharing is possible depending on data safety regulations

REFERENCES:
- [Derived] Schwendner M, Kram L, Zhang H, Krieg SM, Ille S. Preoperative nTMS-based mapping of a verbal semantic association task allows for the identification of extensive bihemispheric cortical and subcortical networks. J Neurooncol. 2025 Dec 8;176(1):108. doi: 10.1007/s11060-025-05355-9. PMID 41359250